CLINICAL TRIAL: NCT03610204
Title: The Effect of Pressure Intensity of a Chinese Massage With the "Buffalo Horn Technique" on Pain Relief for Mechanical Low Back Pain.
Brief Title: Pressure Intensity of a Chinese Massage Technique for Treating Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yen-Nung Lin, Director of Physical Medicine and Rehabilitation, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N201709004
Record Dates: First submitted 2018-07-18; First posted 2018-08-01 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Low Back Pain, Mechanical
Keywords: Alternative therapy; Massage; Manual therapy; Myofascial
MeSH Terms: conditions — Low Back Pain | interventions — Massage

STUDY DESIGN:
Intervention Model Description: The patients are randomly assigned into two treatment arms.
Who Masked: Participant, Outcomes Assessor
Masking Description: Since the patient are prone during the low back massage, the patient will not know what treatment they receive, as the two treatments are similar and only different in the pressure force.
  The primary outcome is assessed by a self-reported questionnaire. The assessor who performs the clinical assessments will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep massage (DM) group (Experimental): The therapist performs the deep massage with "buffalo horn technique". A small rod with a cone-like end was used in the technique. By pressuring the rod end with a higher force against the body surface of the participant, it produces higher pressure that may release the deep-layer fascia of muscles. Thus this technique features a deep massage.
  Interventions: Other: Buffalo horn technique
- Superficial massage (SM) group (Active Comparator): The therapist performs the superficial massage with "buffalo horn technique". By pressuring the rod end with a lower force against the body surface of the participant, it produces lower pressure. Thus this intervention features a superficial massage.
  Interventions: Other: Buffalo horn technique

INTERVENTIONS:
Other: Buffalo horn technique — The participants receive a 30-min massage session, twice a week for a total 6 sessions.
  Other Names: Massage with a Chinese therapeutic tool

SUMMARY:
The Investigators conduct this study to compare two different massage methods with "buffalo horn technique": the deep massage and the superficial massage. To explore the effects of the two interventions on low back pain, the investigators evaluated the outcome measurements regarding pain severity and physical functions before and after 6 times of treatment through a 3-week period.

DETAILED DESCRIPTION:
Background: Nonspecific lower back pain is an important global health issue, with high prevalence over the world and causing huge economic loss.

This research is a double-blind randomized controlled trial. In this study the investigators introduce a technique derived from traditional Chinese massage using a special tool made from buffalo's horns to perform the massage, so called "buffalo horn technique". The tool is like a short rod in about 15-cm length with a cone-like end. During the massage, the therapist presses the cone-like end against the painful region of back. Because the cone-like end has a small contact area with the participant's body surface, it may release deep layer fascia with higher pressure produced by the therapist toward the treatment area. During the intervention of shallow massage, the therapist applies a lower force then that used in the deep massage. Thus it produces a lower pressure on the painful region due to a larger contact surface when pressing the rod end against the body of the participant.

Participants are randomly assigned to either deep-massage group (DM) or superficial-massage (SM) group. The participants received two sessions a week for a total six sessions. The outcome measures include the structured questionnaire to investigate the pain-related outcomes and back pain-related disabilities. The investigators also perform the clinical assessments such as range of motion of trunk. All the outcomes are assessed before-intervention (pretest) and after the end of intervention (posttest).

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Non-specific low back pain over 1 months
3. 20-65 years old
4. No experience of massage therapy within 2 months prior to the study inclusion.

Exclusion Criteria:

1. Pregnancy
2. Back pain associated with systemic disease (autoimmune, infectious, vascular, endocrine, metabolic, or neoplastic disease)
3. Previous spine surgery.
4. Presentation with neurological signs such as radiating pain.
5. .Skin diseases (psoriasis, urticaria, wounds, etc.)

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-26 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) for pain severity | 7 weeks
  0-100mm VAS where 0 represents no pain and 100 represents the strongest pain

SECONDARY OUTCOMES:
Oswestry Disability Index | 7 weeks
  Patients rate the severity (from no problem scored "0" to the worst scored "5") on 10 daily activities. Thus the total scores range from 0 to 50.
Roland-Morris Low Back Pain Disability Questionnaire | 7 weeks
  Participants answer "true" or "false" on 24 items that describe the impact of low back pain on daily activity. Thus the total scores range from 0 to 24.
Short form of "World Health Organization Quality of Life Instrument" (WHOQOL-BREF) | 7 weeks
  The Chinese version has 28 items covering 4 domains in terms of "physical, emotional, social, and environmental". Scores are transformed from 0 to 100 for each domain with higher scores indicating better quality of life.
Pain pressure threshold | 3 weeks
  Using the pressure algometer to measure the pressure enough to elicit the tenderness,
Range of motion (ROM) of the trunk | 3 weeks
  ROM of flexion and extension of the back

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Nung Lin, Principal Investigator — Department of Rehabilitation, Wan-Fang Hospital
Locations (1):
- WanFang Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
only for this study